CLINICAL TRIAL: NCT04749979
Title: Freeze All on Oocyte Maturatin by Gonadotropin Agonist Versus Human Chorionic Gonadotroipin in IVF Cycles
Brief Title: Freeze All on Oocyte Maturatin by Gonadotropin Agonist Versus Human Chorionic Gonadotroipin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Oocyte
Record Dates: First submitted 2021-01-29; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- giving agonist ( eg. decapeptyl ) (Active Comparator): Giving women agonist
  Interventions: Drug: Agonist (decapeptyl )
- Giving HCG (eg. choriomon ) (Active Comparator): Giving women HCG
  Interventions: Drug: HCG ( eg. Choriomon )

INTERVENTIONS:
Drug: Agonist (decapeptyl ) — giving agonist
  Arms: giving agonist ( eg. decapeptyl )
Drug: HCG ( eg. Choriomon ) — giving HCG
  Arms: Giving HCG (eg. choriomon )

SUMMARY:
Estradiol valerate in the form of cycloprogenova™ (white tablet only) was started on day 2 or 3 of cycle with oral dose 4 mg divided on 2 doses in addition to Aspocid 75 mg once daily with folic acid 500 mcg once daily.

DETAILED DESCRIPTION:
U/S was done on day 9 or 10 of cycle to assess endometrial thickness, then every other day until endometrial thickness of 8 mm or more is reached and when endometrial thickness reaches 8 mm or more FET was planned. Progesterone in the form of prontogest™ 400 mg vaginal suppository twice dTwo to Four Day 5 Embryos was transferred

ELIGIBILITY:
Inclusion Criteria:

* PCOS patients according to Rotterdam criteria
* Female age between 20 and 40 years.
* Primary or secondary infertility.
* Body mass index (BMI) between 18 and 40 kg/m2.

Exclusion Criteria:

* Ovarian endometriosis.

  * Ovarian cysts before induction.
  * Known uncontrolled endocrinal abnormalities (like hypo or hyperthyroidism)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females candidate for ICSI
Enrollment: 100 (Estimated)
Dates: Start 2021-02-05 (Estimated); Primary Completion 2021-06-25 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
the number of good quality embryos | within 5 months
  how many good quality embryos

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Principal Investigator — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Aljazeera( Al Gazeera) hospital, Giza, Egypt